CLINICAL TRIAL: NCT06330025
Title: MEasuring and Overcoming Nutritional DIfficulties in Hospitalized Children
Brief Title: Exploring Food Rejection Dispositions as Potential Risk Factors for Undernutrition in Hospitalized Children Aged 2 to 8
Acronym: MEDIALIME
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1180
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Undernutrition
Keywords: Undernutrition; Food intake; Hospitalization; Children; Food rejection; Food neophobia; Food pickiness; Social inequalities
MeSH Terms: conditions — Malnutrition; Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Children between 2 and 8 years, without medical treatments or pathologies impacting food intake and his parents — The group comprises 102 children aged between 2 and 8 years, hospitalized for at least 48 hours and their parents. The children's pathologies and medical treatments should not influence their food intake.

SUMMARY:
Undernutrition affects over 30% of hospitalized children in France, with 10% severely malnourished yet only half of the cases are diagnosed. Undernutrition deteriorates children's health during hospital stays, weakening immunity and hindering recovery. Children suffering from acute malnutrition can stay in the hospital 45% longer than non-malnourished patients.

One of the primary causes of malnutrition is the reduction in children's food intake. Several researchers have emphasized that the young age of patients is associated with reduced food intake. For example, data on 923 children aged 1 day to 16 years indicates that patients under 8 years old are at a higher risk of undernutrition than older children.

The MEDIC project aims to investigate if increased food rejection dispositions contribute to reduced food intake in hospitalized children. Food rejections are typically observed between 2 and 8 years. Some children are more challenging and eat only a few different foods, while others try everything. Around the age of 2, children become more selective about the foods they consume. This is largely due to two common dispositions in young children: food neophobia and food pickiness. Food neophobia is defined as the reluctance to eat or even try foods that appear new, whereas food pickiness is defined as the rejection of a substantial number of familiar foods, including foods previously tasted. Both pickiness and neophobia have been associated with a significant reduction in food consumption (especially of vegetables), a decrease in food variety, and less enjoyment derived from food. A study showed that children aged 2 to 5 were twice as likely to be underweight if they were picky eaters.

Studies have shown that the socioeconomic status has a significant impact on food rejection in children. For instance, longitudinal studies reveal a higher proportion of picky eaters in low-income families. Parental education was also found to be inversely associated with children's food rejection levels.

The MEDIC project seeks to assess health inequalities by studying the impact of food rejection dispositions on the nutritional status of children in pediatric services. A qualitative study supports the notion that food rejection is heightened during the hospitalization: half of the parents of hospitalized children interviewed reported that foods accepted outside the hospital were rejected in the ward. Parents indicated that their child's food preferences were more limited, and they only alternated between a few foods after entering the hospital. According to the majority of interviewed nurses, children refuse any food other than that provided by parents.

The research hypotheses of the MEDIC project focus on understanding the moderating effects of food rejection dispositions and socioeconomic backgrounds on children's food intake during hospitalization. Two hypotheses are formulated: (H1) the pre-hospitalization food rejection levels predict the amount of food consumed during the hospital stay, and (H2) children from disadvantaged socioeconomic backgrounds are more likely to refuse food during their hospital stay than those from more advantaged backgrounds. To test these hypotheses, parents of children aged 2 to 8 will complete questionnaires on food rejection dispositions upon admission, and food consumption (in grams and calories) will be assessed through weighing and photographs of meal trays taken 48 hours (± 24 hours) post-admission. The project aims to shed light on the complexities of childhood malnutrition, addressing social inequalities and contributing valuable insights for interventions and public health policy.

ELIGIBILITY:
Inclusion Criteria:

* child aged between 2 and 8 years (2 years ≤ age ≤ 8 years)
* child admitted to hospitalization for a minimum duration of 48 hours

Exclusion Criteria:

* regularly hospitalized children who come for routine check-ups, thus having repeated exposures to hospital meals
* children with pathologies or treatments causing a significant reduction in their food consumption (perioperative fasting, loss of appetite, nausea, vomiting, etc.)
* children with brain injuries, post-traumatic disorders, sensory deficits, digestive pathologies, severe organ failures (respiratory, cardiac, hepatic, renal)
* children admitted to intensive care units

Ages: 2 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: Study population will include patients between 2 and 8 years admitted to hospitalization for at least 48 hours in a children hospital located in Lyon-France.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Grams of hospital meals consumed by the patients at lunch | Day 2
  To assess the impact of the intensity of food refusal on children's food intake, the investigators will examine the regression coefficient between food refusal scores, measured by the questionnaire completed by one of the patient's parents, and food intake in grams during the lunch 48 hours (± 24 hours) post-admission..
Calories of hospital meals consumed by the patients at lunch, 48 hours after their admission to the hospital. | Day 2
  To assess the impact of the intensity of food refusal on children's food intake, the investigators will examine the regression coefficient between food refusal scores, measured by the questionnaire completed by one of the patient's parents, and food intake in calories during the lunch 48 hours (± 24 hours) post-admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant de Lyon, Bron, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Restier L, Duclos A, Jarri L, Touzet S, Denis A, Occelli P, Kassai-Koupai B, Lachaux A, Loras-Duclaux I, Colin C, Peretti N. Incorrect evaluation of the frequency of malnutrition and of its screening in hospitalized children by health care professionals. J Eval Clin Pract. 2015 Oct;21(5):958-62. doi: 10.1111/jep.12412. Epub 2015 Jul 23. PMID 26202860
- [Background] Joosten KF, Zwart H, Hop WC, Hulst JM. National malnutrition screening days in hospitalised children in The Netherlands. Arch Dis Child. 2010 Feb;95(2):141-5. doi: 10.1136/adc.2008.157255. Epub 2009 May 3. PMID 19414435
- [Background] Mehta NM, Corkins MR, Lyman B, Malone A, Goday PS, Carney LN, Monczka JL, Plogsted SW, Schwenk WF; American Society for Parenteral and Enteral Nutrition Board of Directors. Defining pediatric malnutrition: a paradigm shift toward etiology-related definitions. JPEN J Parenter Enteral Nutr. 2013 Jul;37(4):460-81. doi: 10.1177/0148607113479972. Epub 2013 Mar 25. PMID 23528324
- [Background] Aurangzeb B, Whitten KE, Harrison B, Mitchell M, Kepreotes H, Sidler M, Lemberg DA, Day AS. Prevalence of malnutrition and risk of under-nutrition in hospitalized children. Clin Nutr. 2012 Feb;31(1):35-40. doi: 10.1016/j.clnu.2011.08.011. Epub 2011 Sep 25. PMID 21945311
- [Background] White M, Dennis N, Ramsey R, Barwick K, Graham C, Kane S, Kepreotes H, Queit L, Sweeney A, Winderlich J, Wong See D, Littlewood R. Prevalence of malnutrition, obesity and nutritional risk of Australian paediatric inpatients: a national one-day snapshot. J Paediatr Child Health. 2015 Mar;51(3):314-20. doi: 10.1111/jpc.12709. Epub 2014 Aug 15. PMID 25123425
- [Background] Dovey TM, Staples PA, Gibson EL, Halford JC. Food neophobia and 'picky/fussy' eating in children: a review. Appetite. 2008 Mar-May;50(2-3):181-93. doi: 10.1016/j.appet.2007.09.009. Epub 2007 Sep 29. PMID 17997196
- [Background] Levene IR, Williams A. Fifteen-minute consultation: The healthy child: "My child is a fussy eater!". Arch Dis Child Educ Pract Ed. 2018 Apr;103(2):71-78. doi: 10.1136/archdischild-2016-311787. Epub 2017 Aug 8. PMID 28790134
- [Background] Pliner P, Hobden K. Development of a scale to measure the trait of food neophobia in humans. Appetite. 1992 Oct;19(2):105-20. doi: 10.1016/0195-6663(92)90014-w. PMID 1489209
- [Background] Taylor CM, Wernimont SM, Northstone K, Emmett PM. Picky/fussy eating in children: Review of definitions, assessment, prevalence and dietary intakes. Appetite. 2015 Dec;95:349-59. doi: 10.1016/j.appet.2015.07.026. Epub 2015 Jul 29. PMID 26232139
- [Background] Galloway AT, Lee Y, Birch LL. Predictors and consequences of food neophobia and pickiness in young girls. J Am Diet Assoc. 2003 Jun;103(6):692-8. doi: 10.1053/jada.2003.50134. PMID 12778039
- [Background] Dubois L, Farmer AP, Girard M, Peterson K. Preschool children's eating behaviours are related to dietary adequacy and body weight. Eur J Clin Nutr. 2007 Jul;61(7):846-55. doi: 10.1038/sj.ejcn.1602586. Epub 2006 Dec 20. PMID 17180152
- [Background] Tharner A, Jansen PW, Kiefte-de Jong JC, Moll HA, van der Ende J, Jaddoe VW, Hofman A, Tiemeier H, Franco OH. Toward an operative diagnosis of fussy/picky eating: a latent profile approach in a population-based cohort. Int J Behav Nutr Phys Act. 2014 Feb 10;11:14. doi: 10.1186/1479-5868-11-14. PMID 24512388
- [Background] Vereecken CA, Keukelier E, Maes L. Influence of mother's educational level on food parenting practices and food habits of young children. Appetite. 2004 Aug;43(1):93-103. doi: 10.1016/j.appet.2004.04.002. PMID 15262022
- [Background] Skolin I, Wahlin YB, Broman DA, Koivisto Hursti UK, Vikstrom Larsson M, Hernell O. Altered food intake and taste perception in children with cancer after start of chemotherapy: perspectives of children, parents and nurses. Support Care Cancer. 2006 Apr;14(4):369-78. doi: 10.1007/s00520-005-0904-6. Epub 2006 Jan 28. PMID 16633841